CLINICAL TRIAL: NCT03389763
Title: Comparative Study of Influence of Different Techniques of Remifentanil Titration During Functional Endoscopic Sinus Surgery Under Total Intravenous Anaesthesia (TIVA)
Brief Title: SPI-guided vs PRD-guided Analgesia During FESS for Intraoperative Blood Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Michał Stasiowski, Principal Investigator, 2Department of Anaesthesiology and Intensive Therapy, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SilesianMUKOAiIT3
Record Dates: First submitted 2017-09-06; First posted 2018-01-04 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Endoscopic Sinus Surgery
Keywords: Surgical Pleth Index (SPI); Pupillary Dilatation Reflex (PRD); Intraoperative Blood Loss (IBL); Boezaart Bleeding Scale (BBS); Spectral Entropy (SE); Adequacy of Anaesthesia (AoA); Total Intravenous Anaesthesia (TIVA)
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPI-guided remifentanyl (Experimental): remifentanyl solution will be administered intravenously at a rate 0,25 mcg/kg of body weight/minute, SPI will be monitored on-line; when delta SPI>15, infusion speed of remifentanyl will be increased by 50%
  Interventions: Drug: Remifentanil
- PRD-guided remifentanyl (Experimental): solution remifentanyl solution will be administered intravenously at a rate 0,25 mcg/kg of body weight/minute, PRD measurement every 15 minutes; when PRD>5% infusion speed of remifentanyl will be increased by 50%
  Interventions: Drug: Remifentanil
- BBS-guided remifentanyl (Experimental): BBS assessment every 5 minutes, solution remifentanyl solution will be administered intravenously at a rate 0,25 mcg/kg of body weight/minute; when BBS>2, infusion speed of remifentanyl will be increased by 50%
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — a rate of infusion will be increased by 50% every 5 minutes
  Other Names: Remifentanil infusion

SUMMARY:
The aim of this randomized trial is to assess the efficacy of analgesia , compare the utility of Pupillary Dilatation Reflex (PRD), Surgical Pleth Index (SPI) for monitoring pain perception intraoperatively and their influence on intraoperative blood loss, quality of surgical field using Boezaart Bleeding Scale (BBS) in patients undergoing functional sinus surgery (FESS)

DETAILED DESCRIPTION:
Intraoperative blood loss during FESS constitutes a major problem for a surgeon because it influences quality of surgical field. Each incident of haemorrhage makes the operator stop the procedure in order to bring back the optimal visualization of the intranasal anatomy. In the end it prolongs the time of procedure.

Currently, intraoperative blood loss is estimated based on Boezaart Bleeding Scale (BBS) (0 - no bleeding (cadaveric conditions), 1 - Slight bleeding, no suctioning required, 2 - Slight bleeding, occasional suctioning required, 3 - Slight bleeding, frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed, 4 - Moderate bleeding, frequent suctioning required, and bleeding threatens surgical field directly after suction is removed, 5 - Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible).

Recently, the Surgical Pleth Index (SPI) and Pupillary Dilatation Reflex (PRD) were added as a surrogate variable showing the nociception-antinociception balance into above mentioned parameters constituting a novel approach in monitoring patients intraoperatively, known as adequacy of anaesthesia (AoA) or tailor-made anaesthesia. PRD value >5% reflects increased sensitivity to painful stimulus as well as delta SPI>10 or any SPI>50, and they constitute the indication for administration of rescue analgesia intraoperatively.

This study aims at evaluating utility of SPI-directed analgesia or PRD-directed analgesia or Boezaart scale-directed analgesia using remifentanil on the intraoperative blood loss, haemodynamic stability and time duration of surgery.

Currently, FESS is most often performed using total intravenous anaesthesia (TIVA) which is by majority of anaesthesiologists believed to reduce the intraoperative blood loss compared to general anaesthesia using volatile anaesthetics, but literature provides conflicting findings in this area.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate in the study
* written consent to undergo functional endoscopic sinus surgery under total intravenous anaesthesia
* ASA (American Society of Anesthesiologists) I-III

Exclusion Criteria:

* age under 18 years old
* allergy to propofol
* pregnancy
* any anatomical malformation making PRD or SE measurement impossible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
blood loss postoperatively | end of operation,' assessment
  the investigators will measure the amount of blood loss in the suction bag in millilitres (ml) using a syringe after operation of FESS is completed

SECONDARY OUTCOMES:
heart rate stability intraoperatively | end of operation,' assessment
  the investigators will measure heart rate during TIVAevery 5 minutes up to the end of the operation
hemodynamic stability intraoperatively | intraoperative assessment
  the investigators will measure blood pressure every 5 minutes during TIVA, every 5 minutes up to the end of the operation
PRD-guided pain perception intraoperatively | intraoperative assessment
  The investigators will measure PRD value and adjust infusion speed of remifentanyl, in the case of PRD value >5% the speed of remifentanyl infusion will accelerate by 50%, intraoperatively, every 15 minutes or at any change of BBS, up to the end of the operation
SPI-guided pain perception intraoperatively | intraoperative assessment
  The investigators will measure SPI values and adjust infusion speed of remifentanyl, in the case of delta SPI>15 the speed of remifentanyl infusion will accelerate by 50%, intraoperatively, every 1 minute, up to the end of the operation
condition of surgical field | intraoperative assessment
  the surgeon will assess the quality of surgical field using BBS when the operation of FESS is performed, every 5 minutes or at any change of BBS form the beginning till the end of surgery, up to the end of the operation
total consumption of propofol | end of operation assessment
  The investigators will measure the consumption of propofol intraoperatively
total consumption of remifentanil | end of operation assessment
  The investigators will measure the consumption of remifentanyl intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław O Jałowiecki, Ph.Dr, Principal Investigator — Medical University of Silesia
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
article in Laryngoscope in 2018, case reports
Supporting Information: ICF
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Bhat Pai RV, Badiger S, Sachidananda R, Basappaji SM, Shanbhag R, Rao R. Comparison of surgical conditions following premedication with oral clonidine versus oral diazepam for endoscopic sinus surgery: A randomized, double-blinded study. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):250-6. doi: 10.4103/0970-9185.182112. PMID 27275059
- [Background] Cardesin A, Pontes C, Rosell R, Escamilla Y, Marco J, Escobar MJ, Bernal-Sprekelsen M. Hypotensive anaesthesia and bleeding during endoscopic sinus surgery: an observational study. Eur Arch Otorhinolaryngol. 2014 Jun;271(6):1505-11. doi: 10.1007/s00405-013-2700-0. Epub 2013 Sep 20. PMID 24052249
- [Result] Yoo HS, Han JH, Park SW, Kim KS. Comparison of surgical condition in endoscopic sinus surgery using remifentanil combined with propofol, sevoflurane, or desflurane. Korean J Anesthesiol. 2010 Dec;59(6):377-82. doi: 10.4097/kjae.2010.59.6.377. Epub 2010 Dec 31. PMID 21253373
- [Result] Cafiero T, Cavallo LM, Frangiosa A, Burrelli R, Gargiulo G, Cappabianca P, de Divitiis E. Clinical comparison of remifentanil-sevoflurane vs. remifentanil-propofol for endoscopic endonasal transphenoidal surgery. Eur J Anaesthesiol. 2007 May;24(5):441-6. doi: 10.1017/S0265021506002080. Epub 2007 Mar 12. PMID 17376252
- [Result] Sivaci R, Yilmaz MD, Balci C, Erincler T, Unlu H. Comparison of propofol and sevoflurane anesthesia by means of blood loss during endoscopic sinus surgery. Saudi Med J. 2004 Dec;25(12):1995-8. PMID 15711683
- [Result] Marzban S, Haddadi S, Mahmoudi Nia H, Heidarzadeh A, Nemati S, Naderi Nabi B. Comparison of surgical conditions during propofol or isoflurane anesthesia for endoscopic sinus surgery. Anesth Pain Med. 2013 Sep;3(2):234-8. doi: 10.5812/aapm.9891. Epub 2013 Sep 1. PMID 24282774
- [Result] Cardesin A, Pontes C, Rosell R, Escamilla Y, Marco J, Escobar MJ, Bernal-Sprekelsen M. A randomised double blind clinical trial to compare surgical field bleeding during endoscopic sinus surgery with clonidine-based or remifentanil-based hypotensive anaesthesia. Rhinology. 2015 Jun;53(2):107-15. doi: 10.4193/Rhino14.185. PMID 26030032
- [Result] Drozdowski A, Sieskiewicz A, Siemiatkowski A. [Reduction of intraoperative bleeding during functional endoscopic sinus surgery]. Anestezjol Intens Ter. 2011 Jan-Mar;43(1):45-50. Polish. PMID 21786531
- [Result] Shen PH, Weitzel EK, Lai JT, Wormald PJ, Ho CS. Intravenous esmolol infusion improves surgical fields during sevoflurane-anesthetized endoscopic sinus surgery: a double-blind, randomized, placebo-controlled trial. Am J Rhinol Allergy. 2011 Nov-Dec;25(6):e208-11. doi: 10.2500/ajra.2011.25.3701. PMID 22185726
- [Result] DeConde AS, Thompson CF, Wu EC, Suh JD. Systematic review and meta-analysis of total intravenous anesthesia and endoscopic sinus surgery. Int Forum Allergy Rhinol. 2013 Oct;3(10):848-54. doi: 10.1002/alr.21196. Epub 2013 Jul 10. PMID 23843351
- [Result] Gomez-Rivera F, Cattano D, Ramaswamy U, Patel CB, Altamirano A, Man LX, Luong A, Chen Z, Citardi MJ, Fakhri S. Pilot study comparing total intravenous anesthesia to inhalational anesthesia in endoscopic sinus surgery: novel approach of blood flow quantification. Ann Otol Rhinol Laryngol. 2012 Nov;121(11):725-32. doi: 10.1177/000348941212101105. PMID 23193905
- [Result] Blackwell KE, Ross DA, Kapur P, Calcaterra TC. Propofol for maintenance of general anesthesia: a technique to limit blood loss during endoscopic sinus surgery. Am J Otolaryngol. 1993 Jul-Aug;14(4):262-6. doi: 10.1016/0196-0709(93)90072-f. PMID 8214320
- [Result] Nekhendzy V, Lemmens HJ, Vaughan WC, Hepworth EJ, Chiu AG, Church CA, Brock-Utne JG. The effect of deliberate hypercapnia and hypocapnia on intraoperative blood loss and quality of surgical field during functional endoscopic sinus surgery. Anesth Analg. 2007 Nov;105(5):1404-9, table of contents. doi: 10.1213/01.ane.0000282781.56025.52. PMID 17959973
- [Result] Manola M, De Luca E, Moscillo L, Mastella A. Using remifentanil and sufentanil in functional endoscopic sinus surgery to improve surgical conditions. ORL J Otorhinolaryngol Relat Spec. 2005;67(2):83-6. doi: 10.1159/000084576. Epub 2005 Mar 22. PMID 15785115
- [Result] Puthenveettil N, Rajan S, Kumar L, Nair SG. A comparison of effects of oral premedication with clonidine and metoprolol on intraoperative hemodynamics and surgical conditions during functional endoscopic sinus surgery. Anesth Essays Res. 2013 Sep-Dec;7(3):371-5. doi: 10.4103/0259-1162.123244. PMID 25885986
- [Result] Guglielminotti J, Grillot N, Paule M, Mentre F, Servin F, Montravers P, Longrois D. Prediction of movement to surgical stimulation by the pupillary dilatation reflex amplitude evoked by a standardized noxious test. Anesthesiology. 2015 May;122(5):985-93. doi: 10.1097/ALN.0000000000000624. PMID 25730338
- [Result] Paulus J, Roquilly A, Beloeil H, Theraud J, Asehnoune K, Lejus C. Pupillary reflex measurement predicts insufficient analgesia before endotracheal suctioning in critically ill patients. Crit Care. 2013 Jul 24;17(4):R161. doi: 10.1186/cc12840. PMID 23883683
- [Result] Migeon A, Desgranges FP, Chassard D, Blaise BJ, De Queiroz M, Stewart A, Cejka JC, Combet S, Rhondali O. Pupillary reflex dilatation and analgesia nociception index monitoring to assess the effectiveness of regional anesthesia in children anesthetised with sevoflurane. Paediatr Anaesth. 2013 Dec;23(12):1160-5. doi: 10.1111/pan.12243. Epub 2013 Aug 2. PMID 23910160
- [Result] Aissou M, Snauwaert A, Dupuis C, Atchabahian A, Aubrun F, Beaussier M. Objective assessment of the immediate postoperative analgesia using pupillary reflex measurement: a prospective and observational study. Anesthesiology. 2012 May;116(5):1006-12. doi: 10.1097/ALN.0b013e318251d1fb. PMID 22446982